CLINICAL TRIAL: NCT05814198
Title: Evaluation of Hemoglobin, Albumin, Lymphocyte, Platelet (HALP) Score in Distinction Between Fetal Growth Restriction (FGR) and Small for Gestational Age (SGA)
Brief Title: Evaluation of HALP Score in Distinction Between FGR and SGA
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, murat ibrahim toplu, medical doctor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 78
Record Dates: First submitted 2023-04-01; First posted 2023-04-14 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Fetal Growth Restriction; Small for Gestational Age at Delivery
Keywords: fetal growth restriction; small for gestational age
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FGR: In the group with FGR, we will calculate the HALP score with the complete blood count and albumin values.
  Interventions: Diagnostic Test: HALP score
- SGA: In the group with SGA, we will calculate the HALP score with the complete blood count and albumin values.
  Interventions: Diagnostic Test: HALP score

INTERVENTIONS:
Diagnostic Test: HALP score — we will calculate the HALP score with the complete blood count and albumin values in FGR and SGA groups.

SUMMARY:
Fetal Growth Restriction (FGR) and Small for Gestational Age (SGA) are two conditions that can happen when a baby doesn't grow as much as expected during pregnancy. FGR is caused by things like problems with the mother's nutrition and inflammation, while SGA is usually because of genetic and other factors.

It's important to know if a baby has FGR or SGA because FGR babies can have more health problems and are at risk of dying before or shortly after birth. SGA babies are usually healthy, but they might have more health problems later in life.

Doctors can use a simple blood test called the HALP score to see if a mother has problems with her nutrition and inflammation. However, it hasn't been studied for FGR and SGA. We want to study if the HALP score can help us tell if a baby has FGR or SGA by looking at the mother's blood test results.

DETAILED DESCRIPTION:
Fetal Growth Restriction (FGR) and Small for Gestational Age (SGA) are two conditions that are commonly encountered in obstetrics. FGR is defined as a condition in which the fetus is smaller than expected for its gestational age, and its pathophysiology is thought to be influenced by both maternal inflammation and nutritional status. On the other hand, SGA is a condition in which the fetus is smaller than expected, but its pathophysiology is primarily attributed to constitutional and genetic factors.

It is important to distinguish between FGR and SGA because FGR is associated with a higher risk of adverse fetal and neonatal outcomes, including morbidity and mortality. In contrast, SGA infants are generally healthy, but may have a higher risk of long-term health problems, such as hypertension and diabetes.

The HALP score is a simple and easily calculated index that is based on the levels of hemoglobin, lymphocytes, albumin, and platelets. It has been shown to be informative about the nutritional and inflammatory status in various medical fields. However, its use in obstetrics is limited and its potential to distinguish between FGR and SGA has not been studied.

Given that maternal inflammation and nutritional status are also involved in the pathophysiology of FGR, it is possible that the HALP score could be useful in distinguishing between FGR and SGA. Therefore, we plan to investigate the potential of the HALP score in differentiating between these two conditions.

ELIGIBILITY:
Inclusion Criteria:

* Having a singleton pregnancy
* Pregnant women diagnosed with FGR and SGA in accordance with the criteria of the International Society of Ultrasound in Obstetrics and Gynecology (ISUOG) diagnosis and management bulletin in SGA and FGR
* Pregnant women who do not have a systemic inflammatory disease other than FGR
* Pregnant women whose delivery and postpartum follow-up are in our clinic
* Pregnant women who have no history or signs of systemic disease
* Pregnant women who have not found any maternal or fetal abnormality in the pregnancy follow-up

Exclusion Criteria:

* Multiple gestation pregnancies
* Known chronic or systemic disease (hypo or hyperthyroidism, diabetes, chronic hypertension, heart diseases, hyperlipidemia, chronic liver failure, acute or chronic kidney failure, etc.)
* Pregnant women whose pregnancy follow-up is unknown or fetal or maternal abnormalities are detected in the follow-up
* Pregnant women whose delivery or postpartum follow-up is in a location other than our clinic

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women between the ages of 18-44 who were diagnosed with FGR and SGA in our clinic and whose follow-up and birth were in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Evaluate Hemoglobin, Albumin, Lymphocyte, and Platelet (HALP) Score in Fetal Growth Restriction (FGR) and Small for Gestational Age (SGA) groups | Data assessed from patient charts retrospectively/From January 2021 to January 2023, pregnant women who are diagnosed with FGR and SGA, will have their examination findings and medical tests documented by scanning patient records.
  The Hemoglobin, Albumin, Lymphocyte, Platelet (HALP) score represents a valuable tool for clinicians to assess a patient's nutritional and inflammatory status. Elevated HALP scores are indicative of superior immune-nutritional function, while lower scores are suggestive of poorer immune-nutritional status. As such, the HALP score offers important prognostic information that may inform treatment decisions and risk stratification for patients with various medical conditions. There is no standardized or universal threshold for the HALP score to stratify the risk of these outcomes. Based on the existing literature, the meaningful cutoff for HALP is disease-specific and largely study-specific.

CONTACTS AND LOCATIONS:
Overall Officials: murat i toplu, MD, Principal Investigator — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Locations (1):
- Prof. Dr. Cemil Taşcıoğlu City Hospital, Istanbul, Turkey (Türkiye)